CLINICAL TRIAL: NCT02643368
Title: Assessing Immunogenicity of Type 2 Monovalent Oral Poliovirus Vaccine Administered at One, Two or Four Week Intervals and When Coadministered With Inactivated Poliovirus Vaccine in an Urban Area in Bangladesh
Brief Title: Immunogenicity of Monovalent Type 2 Oral Poliovirus Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ICDDRB-RRC-PR-15085
Record Dates: First submitted 2015-12-10; First posted 2015-12-31 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2016-03

CONDITIONS: Poliomyelitis
Keywords: Polio; Inactivated polio vaccine; oral polio vaccine; monovalent type 2 oral polio vaccine
MeSH Terms: conditions — Poliomyelitis | interventions — Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- mOPV2 at 6 and 7 weeks of age (Active Comparator): Participants enrolled in this arm would receive a dose of monovalent type 2 oral polio vaccine (mOPV2) at 6 and 7 weeks of age
  Interventions: Biological: mOPV2 at 6 and 7 weeks of age
- mOPV2 at 6 and 8 weeks of age (Active Comparator): Participants enrolled in this arm would receive a dose of monovalent type 2 oral polio vaccine (mOPV2) at 6 and 8 weeks of age
  Interventions: Biological: mOPV2 at 6 and 8 weeks of age
- mOPV2 at 6 and 10 weeks of age (Active Comparator): Participants enrolled in this arm would receive a dose of monovalent type 2 oral polio vaccine (mOPV2) at 6 and 10 weeks of age
  Interventions: Biological: mOPV2 at 6 and 10 weeks of age
- mOPV2 at 6 and 10 week of age and IPV at 6 weeks of age (Active Comparator): Participants enrolled in this arm would receive a dose monovalent type 2 oral polio vaccine (mOPV2) at 6 and 10 weeks of age. In addition, the participants will also receive inactivated polio vaccine (IPV) at 6 weeks of age
  Interventions: Biological: mOPV2 at 6 and 10 weeks of age; Biological: IPV at 6 weeks of age

INTERVENTIONS:
Biological: mOPV2 at 6 and 7 weeks of age — Participants assigned to this intervention will receive a dose of monovalent oral type 2 polio vaccine (mOPV2) at 6 and 7 weeks of age
  Arms: mOPV2 at 6 and 7 weeks of age
Biological: mOPV2 at 6 and 8 weeks of age — Participants assigned to this intervention will receive a dose of monovalent oral type 2 polio vaccine (mOPV2) at 6 and 8 weeks of age
  Arms: mOPV2 at 6 and 8 weeks of age
Biological: mOPV2 at 6 and 10 weeks of age — Participants assigned to this intervention will receive a dose of monovalent oral type 2 polio vaccine (mOPV2) at 6 and 10 weeks of age
  Arms: mOPV2 at 6 and 10 week of age and IPV at 6 weeks of age; mOPV2 at 6 and 10 weeks of age
Biological: IPV at 6 weeks of age — Participants assigned to this intervention will receive a dose of inactivated polio vaccine (IPV) 6 weeks of age
  Arms: mOPV2 at 6 and 10 week of age and IPV at 6 weeks of age

SUMMARY:
This is an open-label phase IV, randomized controlled trial of mOPV2 alone and mOPV2 along with IPV. This trial will assess the impact on type 2 immunogenicity by reducing the interval between mOPV2 doses. The trial will also evaluate any difference in immunogenicity when the first dose of mOPV2, in a two dose schedule with a four week interval, is administered simultaneously with IPV.

DETAILED DESCRIPTION:
The Strategic Advisory Group of Experts on Immunization (SAGE) has recommended a phased cessation of OPVs starting with serotype 2 (OPV2). This is because the last case of type 2 wild poliovirus (WPV2) was reported in 1999 and type 2 vaccine poliovirus is associated with the highest risk of causing paralysis due to reversion to vaccine derived poliovirus (VDPV), in which the reverted virus acquires not only the ability to cause paralysis but also the ability to transmit from person-to-person. Withdrawal of OPV2 will be done through the replacement worldwide of trivalent OPV (tOPV) with bivalent (types 1 and 3) OPV (bOPV) for use in routine immunization and in campaigns.

After the tOPV to bOPV switch, there will be strict biosafety requirements for the use of vaccines containing OPV2. Trivalent OPV will no longer exist and use of monovalent OPV2 (mOPV2) will be limited to responding to a type 2 outbreak. To respond to poliovirus type 2 outbreaks, the Global Polio Eradication Initiative has proposed delivering using mOPV2 in campaigns conducted in the primary zone of the outbreak and IPV in campaigns conducted in areas adjacent to outbreak zone. Therefore, mOPV2 will be a critical component of response to poliovirus type 2 outbreaks.

Typically, polio campaigns are conducted at an interval of 4 weeks. Recently, a clinical trial conducted by icddr,b and the U.S. Centers for Disease Control and Prevention (CDC) in Matlab and Mirpur in Bangladesh demonstrated non-inferiority of type 1 seroconversion after bOPV or mOPV1 at a 2 week interval compared to 4 weeks between doses. Based these findings, the Global Polio Eradication Initiative (GPEI) concluded that the immune response to "OPV is satisfactory when the interval between doses is shortened to 14 or even 7 days (in case of mOPV1)" and has used short-interval campaigns to deliver mOPV1 and bOPV in areas with security-limited access and for outbreak response. However, there are no data and no current or planned polio clinical trials are assessing the impact on immunogenicity of mOPV2 of a reduction in the interval between mOPV2 doses or of administration of mOPV2 in combination with IPV. Therefore, the findings from the trial proposed in this protocol have a direct and immediate implication on strategies to respond to type 2 polio outbreaks.

Field site: The study will be carried out in urban slums in Mirpur and Mohakahli in Dhaka.

ELIGIBILITY:
Inclusion Criteria:

* Infants 6 weeks of age (range: 42-48 days).
* Parents that consent for participation in the full length of the study.
* Parents that are able to understand and comply with planned study procedures.

Exclusion Criteria:

* Parents and infants who are unable to participate in the full length of the study.
* Evidence of a chronic medical condition identified during physical exam.
* A diagnosis or suspicion of immunodeficiency disorder either in the infant or in an immediate family member.
* A diagnosis or suspicion of bleeding disorder that would contraindicate parenteral administration of IPV or collection of blood by venipuncture.
* Acute diarrhea, infection or illness at the time of enrollment (6 weeks of age) that would require infant's admission to a hospital or would contraindicate provision of OPV or IPV per country guidelines.
* Acute vomiting and intolerance to liquids within 24 hours before the enrollment visit (6 weeks of age).
* Receipt of any polio vaccine (OPV or IPV) before enrollment based upon documentation or parental recall.
* Known allergy/sensitivity or reaction to polio vaccine or contents of polio vaccine.
* Infants from multiple births. Infants from multiple births will be excluded to reduce the potential for contact transmission of vaccine poliovirus to siblings. The infant(s) from a multiple birth who is/are not enrolled would be likely to receive routine immunization and transmit vaccine poliovirus to the enrolled infant.
* Infants from premature births (<37 weeks of gestation).

Ages: 6 Weeks to 7 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 760 (Actual)
Dates: Start 2015-12; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Assessment of type 2 immunogenicity | The antibody titers 4 weeks after completing the vaccination schedule compared to that at 6 weeks of age.
  To assess type 2 immunogenicity seroconversion will be determined in each study arm. Seroconversion will be defined as either a four-fold increase from the titer predicted after accounting for the expected decline in maternal antibodies, assuming a half-life of 28 days, or a seronegative participant (<1:8 titers) who becomes seropositive (≥1:8). The antibody titers at 6 weeks of age will be assumed to be the starting point for the expected decline in maternal antibody. The endpoint titer assessment will be 4 weeks after completing study vaccination schedule.

CONTACTS AND LOCATIONS:
Locations (1):
- International Center for Diarrhoeal Disease Research, Bangladesh, Dhaka, Bangladesh

REFERENCES:
- [Derived] Zaman K, Estivariz CF, Morales M, Yunus M, Snider CJ, Gary HE Jr, Weldon WC, Oberste MS, Wassilak SG, Pallansch MA, Anand A. Immunogenicity of type 2 monovalent oral and inactivated poliovirus vaccines for type 2 poliovirus outbreak response: an open-label, randomised controlled trial. Lancet Infect Dis. 2018 Jun;18(6):657-665. doi: 10.1016/S1473-3099(18)30113-0. Epub 2018 Mar 20. PMID 29571817